CLINICAL TRIAL: NCT01025882
Title: Phase I Study of Margin-Intense Combination Therapy for Patients With Potentially Resectable Pancreatic Adenocarcinoma
Brief Title: Margin-Intense Combo Therapy in Pts w/Potentially Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: DSMC closed due to patient deaths
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-01209; CDR0000657523 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01117 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Regimen 1 (Experimental): Patients undergo a single fraction of margin-intensive stereotactic body radiotherapy (SBRT) on day 1. Patients undergo pancreatoduodenectomy between days 15-43.
  Interventions: Radiation: stereotactic body radiation therapy
- Regimen 2 (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients undergo a single fraction of SBRT between days 21-28 followed by pancreatoduodenectomy between days 35-63.
  Interventions: Drug: gemcitabine hydrochloride; Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Arms: Regimen 2
Radiation: stereotactic body radiation therapy — Given as a single fraction

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving stereotactic body radiation therapy together with gemcitabine hydrochloride may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of stereotactic body radiation therapy when given with or without gemcitabine hydrochloride in treating patients with pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To demonstrate the feasibility and safety of administering margin-intensive stereotactic body radiotherapy together with preoperative gemcitabine hydrochloride to patients with resectable pancreatic adenocarcinoma.

OUTLINE: This is a multicenter, dose-escalation study of gemcitabine hydrochloride. Patients receive 1 of 2 treatment regimens.

* Regimen 1: Patients undergo a single fraction of margin-intensive stereotactic body radiotherapy (SBRT) on day 1. Patients undergo pancreatoduodenectomy between days 15-43.
* Regimen 2: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients undergo a single fraction of SBRT between days 21-28 followed by pancreatoduodenectomy between days 35-63.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed localized adenocarcinoma of the pancreas or distal common bile duct

  * Pancreatic ductal adenocarcinoma or peripancreatic cholangiocarcinoma
* Resectable disease, as determined by the Gastrointestinal Cancer Working Group disease-oriented team

  * Criteria used to define unresectability will include, but not be limited to, the following:

    * Tumor encases > 180 degrees of the circumference of the superior mesenteric artery
    * Tumor encases the common hepatic artery with no anatomic option for reconstruction following segmental resection
    * Superior mesenteric vein occluded or encased with no option for reconstruction following segmental resection
    * Soft tissue infiltration of the retroperitoneum to the left of the superior mesenteric artery
* All malignant disease must be encompassed within a single radiotherapy field
* No metastatic disease

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute granulocyte count > 1,500/mm³
* Platelet count > 100,000/mm³
* Creatinine clearance > 50mL/min
* AST and ALT < 5 times upper limit of normal
* Serum bilirubin < 5 mg/dL (with biliary decompression)
* INR ≤ 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Medically fit for pancreatic surgical resection, as determined by the investigating surgeons at the time of study enrollment
* No evidence of an active second invasive malignancy outside the area of the pancreas or biliary system within the past 2 years, except for non-melanomatous skin cancer or carcinoma in situ of the breast, bladder, cervix, or uterus
* No clinically significant cardiac disease, including the following:

  * Uncontrolled hypertension, defined as blood pressure > 160/90 mm Hg on medication
  * Myocardial infarction within the past 6 months
  * NYHA class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication (e.g., chronic atrial arrhythmia [atrial fibrillation or paroxysmal supraventricular tachycardia])

    * Atrial arrhythmia allowed provided it is well-controlled on stable medication
  * No current or recent (within the past 6 months) unstable angina
* No recent (within the past 6 months) arterial thromboembolic events, including transient ischemic attack, cerebrovascular accident, or clinically significant peripheral artery disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No serious nonhealing wound, ulcer, or currently healing fracture
* No AIDS
* No significant infection or other coexisting medical condition that would preclude study therapy
* No gastrointestinal fistula or perforation within the past 10 years

PRIOR CONCURRENT THERAPY:

* More than 2 years since prior chemotherapy (other than for pancreaticobiliary cancer)
* More than 28 days since prior major surgical procedure or open biopsy
* No prior intraabdominal radiotherapy in the planned field of pancreatic margin-intensive radiotherapy
* No prior organ transplantation
* No concurrent major surgical procedure
* No other concurrent cytotoxic chemotherapy or anti-neoplastic biologic agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02-18 (Actual); Study Completion 2011-02-18 (Actual)

PRIMARY OUTCOMES:
Preoperative treatment-related toxicity, defined as adverse events occurring prior to surgical resection
Postoperative surgical morbidity, defined as all other adverse events occurring within 90 days of surgery
Total dose of chemotherapy and radiotherapy delivered
Pre-treatment and post-treatment characteristics of the primary tumor on preoperative axial imaging including, but not limited to, tumor size, percentage of encasement/abutment of mesenteric vessels, and progression of disease
Postoperative complications including, but not limited to, need for reoperation, need for interventional radiology fluid collection drainage, systemic infection, wound infection, prolonged ICU stay, and delayed gastric emptying
Operative drain amylase at days 3 and 5 postoperatively
Length of hospital stay following pancreatic resection
Degree of histologic response of tumor in the resected specimen
Tumor samples for RNA and protein harvesting (when possible) from pretreatment biopsies and surgical specimens

CONTACTS AND LOCATIONS:
Overall Officials: John C. Mansour, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States